CLINICAL TRIAL: NCT05434273
Title: The Effects of an Integrated Exercise and Cardiovascular Health Education Programme on Community-dwelling Older Adults at Risk of Atherosclerotic Cardiovascular Diseases: A Randomised Controlled Trial
Brief Title: Effects of Integrated Cardiovascular Health Education Program on Older Adults at Risk of ASCVD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Eva Ho, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ASCVD_OlderAdult_Full
Record Dates: First submitted 2022-06-11; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Cardiovascular Diseases; Healthy Lifestyle; Health Education
Keywords: Older Adults; Physical Activity; Atherosclerotic Cardiovascular Disease; Lifestyle Modification; Health Education
MeSH Terms: conditions — Cardiovascular Diseases; Health Education; Motor Activity; Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm: Integrated Intervention (Experimental): Receive an integrated exercise and cardiovascular health education programme (HE programme)
  Interventions: Behavioral: HE programme
- Control (Sham Comparator): Receive usual care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: HE programme — Participants will receive a 12-week integrated exercise and cardiovascular health education programme (HE programme) which is constructed based on self-efficacy theory. A booster intervention in the form of SMS messaging will be given from Week 1 to Week 12.
  Arms: Experimental Arm: Integrated Intervention
Behavioral: Usual care — Participants will receive usual care which primarily includes an education talk on basic health issues. A governmental health education leaflet and a lecture video will be provided for reference.
  Arms: Control

SUMMARY:
Despite older adults being exposed to an increased risk of atherosclerotic cardiovascular disease (ASCVD), they are generally underrepresented in cardiovascular prevention programmes. The aim of this study is to examine the effects of an integrated exercise and cardiovascular health education programme (HE programme) on community-dwelling older adults at risk of ASCVD.

DETAILED DESCRIPTION:
The study is a two-arm randomized controlled trial. (1) The control group will mainly receive a basic lifestyle modification talk, a lecture video and governmental education leaflets. (2) The experimental group will receive an integrated exercise and health education programme (HE programme) based on self-efficacy theory. Physical activity level, exercise self-efficacy and ASCVD risk profile including blood pressure, cardiac endurance, fasting blood glucose, fasting blood lipids, and anthropometric outcomes will be investigated via physiological assessments, medical history-taking or questionnaires at baseline, Week 12, Week 24 and Week 36.

ELIGIBILITY:
Inclusion Criteria:

* Chinese adults ≧60 years old
* Having at least one ASCVD risk factor
* Pass the cardiovascular fitness evaluation
* Able to write and read Chinese, and communicate in Cantonese;
* Possess a mobile phone and able to make use of the phone in reading short messages

Exclusion Criteria:

* Visually impaired, hearing impaired, or suffer from cognitive, psychiatric, or muscular disorder
* Having a history of attending similar cardiovascular prevention program
* Having a previous history of coronary heart disease or stroke

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Physical activity level (total score) at Week 24 | At Week 24
  The physical activity level will be measured by the Chinese Version of Physical Activity Scale for the Elderly (PASE-C). The total score (from zero to 400 or above) is quantified based on frequency values and weights for these activities. The higher the score, the higher the level of physical activity.
Physical activity level (classification of physical activity level) at Week 24 | At Week 24
  The physical activity level will be measured by the Chinese version of International Physical Activity Questionnaire-short form (IPAQ-C-short form). Participants are classified into "inactive", "minimally active" or "health enhancing physical activity (HEPA) active" based on their physical activity levels.

SECONDARY OUTCOMES:
Exercise self-efficacy at baseline | At baseline
  Exercise self-efficacy will be measured via the Chinese version of Self-Efficacy for Exercise (SEE-C). The total score ranges from 0 to 90. The higher the score, the greater the exercise self-efficacy.
Exercise self-efficacy at Week 12 | At Week 12
  Exercise self-efficacy will be measured via the Chinese version of Self-Efficacy for Exercise (SEE-C). The total score ranges from 0 to 90. The higher the score, the greater the exercise self-efficacy.
Exercise self-efficacy at Week 24 | At Week 24
  Exercise self-efficacy will be measured via the Chinese version of Self-Efficacy for Exercise (SEE-C). The total score ranges from 0 to 90. The higher the score, the greater the exercise self-efficacy.
Exercise self-efficacy at Week 36 | At Week 36
  Exercise self-efficacy will be measured via the Chinese version of Self-Efficacy for Exercise (SEE-C). The total score ranges from 0 to 90. The higher the score, the greater the exercise self-efficacy.
ASCVD risk profiles (Blood pressure, weight, height, BMI & waist circumference, heart rate) at baseline | At baseline
  The ASCVD risk profiles will be assessed by physical evaluations carried out by blinded, trained outcome assessors.
ASCVD risk profiles (Blood pressure, weight, height, BMI & waist circumference, heart rate) at Week 12 | At Week 12
  The ASCVD risk profiles will be assessed by physical evaluations carried out by blinded, trained outcome assessors.
ASCVD risk profiles (Blood pressure, weight, height, BMI & waist circumference, heart rate) at Week 24 | At Week 24
  The ASCVD risk profiles will be assessed by physical evaluations carried out by blinded, trained outcome assessors.
ASCVD risk profiles (Blood pressure, weight, height, BMI & waist circumference, heart rate) at Week 36 | At Week 36
  The ASCVD risk profiles will be assessed by physical evaluations carried out by blinded, trained outcome assessors.
ASCVD risk profiles (Fasting blood glucose and fasting blood lipids including low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL) cholesterol, and triglycerides) at baseline | At baseline
  The ASCVD risk profiles will be assessed by obtaining finger-prick blood samples using an auto-analyser, carried out by blinded, trained outcome assessors. Fasting 8 hours before obtaining blood samples will be required.
ASCVD risk profiles (Fasting blood glucose and fasting blood lipids including low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL) cholesterol, and triglycerides) at Week 24 | At Week 24
  The ASCVD risk profiles will be assessed by obtaining finger-prick blood samples using an auto-analyser, carried out by blinded, trained outcome assessors. Fasting 8 hours before obtaining blood samples will be required.
ASCVD risk profiles (Fasting blood glucose and fasting blood lipids including low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL) cholesterol, and triglycerides) at Week 36 | At Week 36
  The ASCVD risk profiles will be assessed by obtaining finger-prick blood samples using an auto-analyser, carried out by blinded, trained outcome assessors. Fasting 8 hours before obtaining blood samples will be required.
ASCVD risk profiles (2-minute walk test) at baseline | At baseline
  2-minute walk test will be adopted to examine aerobic capacity and self-paced walking capacity by measuring the walking distance covered at two minutes. It will be assessed by blinded, trained outcome assessors.
ASCVD risk profiles (2-minute walk test) at Week 12 | At Week 12
  2-minute walk test will be adopted to examine aerobic capacity and self-paced walking capacity by measuring the walking distance covered at two minutes. It will be assessed by blinded, trained outcome assessors.
ASCVD risk profiles (2-minute walk test) at Week 24 | At Week 24
  2-minute walk test will be adopted to examine aerobic capacity and self-paced walking capacity by measuring the walking distance covered at two minutes. It will be assessed by blinded, trained outcome assessors.
ASCVD risk profiles (2-minute walk test) at Week 36 | At Week 36
  2-minute walk test will be adopted to examine aerobic capacity and self-paced walking capacity by measuring the walking distance covered at two minutes. It will be assessed by blinded, trained outcome assessors.
Adverse events throughout the program | Throughout the study period
  Unfavorable or unintended events regarding the programme reported by participants throughout the study period.
Eligibility rate | At baseline
  The number of eligible potential participants divided by the number of screened people
Recruitment rate | At baseline
  The percentage of participants who consent to join the study and being recruited
Retention rate at baseline | At baseline
  The percentage of participants remaining in the study
Retention rate at Week 12 | At Week 12
  The percentage of participants remaining in the study
Retention rate at Week 24 | At Week 24
  The percentage of participants remaining in the study
Retention rate at Week 36 | At Week 36
  The percentage of participants remaining in the study
Lecture attendance rate | Immediately after education session
  The number of participants in the control group who attend the education talk divided by the number of participants who are randomized into the control group The number of participants in the experimental group who attend the education session divided by the number of participants who are randomized into the experimental group The number of participants in the two groups who attend the education session divided by the number of randomized participants
Adherence to intervention | At Week 36
  The number of participants in the experimental group who practice the tailor-made exercise learned during the intervention divided by the number of participants in the experimental group Experimental group's frequency in performing tailor-made exercise related to the recommended exercise dosage
Attendance rate to data collection at baseline | At baseline
  The number of participants in the control group who attend the data collection divided by the number of participants who are randomized into the control group The number of participants in the experimental group who attend the data collection divided by the number of participants who are randomized into the experimental group The number of participants who attend the data collection divided by the number of randomized participants
Attendance rate to data collection at Week 12 | At Week 12
  The number of participants in the control group who attend the data collection divided by the number of participants who are randomized into the control group The number of participants in the experimental group who attend the data collection divided by the number of participants who are randomized into the experimental group The number of participants who attend the data collection divided by the number of randomized participants
Attendance rate to data collection at Week 24 | At Week 24
  The number of participants in the control group who attend the data collection divided by the number of participants who are randomized into the control group The number of participants in the experimental group who attend the data collection divided by the number of participants who are randomized into the experimental group The number of participants who attend the data collection divided by the number of randomized participants
Attendance rate to data collection at Week 36 | At Week 36
  The number of participants in the control group who attend the data collection divided by the number of participants who are randomized into the control group The number of participants in the experimental group who attend the data collection divided by the number of participants who are randomized into the experimental group The number of participants who attend the data collection divided by the number of randomized participants
Questionnaire completion rate at baseline | At baseline
  The number of participants who complete the questionnaire divided by the number of distributed questionnaires
Questionnaire completion rate at Week 12 | At Week 12
  The number of participants who complete the questionnaire divided by the number of distributed questionnaires
Questionnaire completion rate at Week 24 | At Week 24
  The number of participants who complete the questionnaire divided by the number of distributed questionnaires
Questionnaire completion rate at Week 36 | At Week 36
  The number of participants who complete the questionnaire divided by the number of distributed questionnaires
Missing data at baseline | At baseline
  The percentage of missing data
Missing data at Week 12 | At Week 12
  The percentage of missing data
Missing data at Week 24 | At Week 24
  The percentage of missing data
Missing data at Week 36 | At Week 36
  The percentage of missing data
Structured questionnaire | At baseline
  The questionnaire will primarily include patient demographics, medical history, lifestyle patterns, medication use and physical fitness evaluation data, etc.
Physical activity level (total score) at baseline | At baseline
  The physical activity level will be measured by the Chinese Version of Physical Activity Scale for the Elderly (PASE-C). The total score (from zero to 400 or above) is quantified based on frequency values and weights for these activities. The higher the score, the higher the level of physical activity.
Physical activity level (total score) at Week 12 | At Week 12
  The physical activity level will be measured by the Chinese Version of Physical Activity Scale for the Elderly (PASE-C). The total score (from zero to 400 or above) is quantified based on frequency values and weights for these activities. The higher the score, the higher the level of physical activity.
Physical activity level (total score) at Week 36 | At Week 36
  The physical activity level will be measured by the Chinese Version of Physical Activity Scale for the Elderly (PASE-C). The total score (from zero to 400 or above) is quantified based on frequency values and weights for these activities. The higher the score, the higher the level of physical activity.
Physical activity level (classification of physical activity level) at baseline | At baseline
  The physical activity level will be measured by the Chinese version of International Physical Activity Questionnaire-short form (IPAQ-C-short form). Participants are classified into "inactive", "minimally active" or "health enhancing physical activity (HEPA) active" based on their physical activity levels.
Physical activity level (classification of physical activity level) at Week 12 | At Week 12
  The physical activity level will be measured by the Chinese version of International Physical Activity Questionnaire-short form (IPAQ-C-short form). Participants are classified into "inactive", "minimally active" or "health enhancing physical activity (HEPA) active" based on their physical activity levels.
Physical activity level (classification of physical activity level) at Week 36 | At Week 36
  The physical activity level will be measured by the Chinese version of International Physical Activity Questionnaire-short form (IPAQ-C-short form). Participants are classified into "inactive", "minimally active" or "health enhancing physical activity (HEPA) active" based on their physical activity levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yan Ho, Study Director — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Lo FMW, Wong EML, Ho KY. The effects of an integrated exercise and cardiovascular health education programme on community-dwelling older adults at risk of atherosclerotic cardiovascular diseases: A study protocol for a randomised controlled trial. PLoS One. 2023 May 24;18(5):e0286181. doi: 10.1371/journal.pone.0286181. eCollection 2023. PMID 37224162